CLINICAL TRIAL: NCT02351687
Title: Randomized Controlled Trial of the Impact of Offering a Nutrition and Health Intervention to Children Recovered From Moderate Acute Malnutrition
Brief Title: Package of Interventions After Recovering From Moderate Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFU2014
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Malnutrition
Keywords: Moderate Acute Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — fanasil, pyrimethamine drug combination; Albendazole; Zinc; Insecticide-Treated Bednets

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention (No Intervention): No specific intervention given after recovery from moderate acute malnutrition.
- Package of interventions (Experimental): Package of interventions given after recovery from moderate acute malnutrition -- includes lipid-nutrient supplement for 2 months, malaria chemoprophylaxis for 3 months during malaria season, an insecticide-treated bed net, a one-time albendazole treatment, and 14 days of zinc.
  Interventions: Dietary Supplement: Lipid Nutrient Supplement; Drug: Sulfadoxine-pyrimethamine; Drug: Albendazole; Drug: Zinc; Other: Insecticide-treated bednet

INTERVENTIONS:
Dietary Supplement: Lipid Nutrient Supplement
  Arms: Package of interventions
Drug: Sulfadoxine-pyrimethamine
  Arms: Package of interventions
Drug: Albendazole
  Arms: Package of interventions
Drug: Zinc
  Arms: Package of interventions
Other: Insecticide-treated bednet
  Arms: Package of interventions

SUMMARY:
Children who recover from moderate acute malnutrition in Malawi remain at high risk for relapse or death in the year following recovery. This cluster-randomized trial will evaluate a package of affordable, safe, proven interventions specifically targeted to this population of children in an attempt to decrease their risk of relapse or death following recovery from moderate acute malnutrition. These children will be followed for a year following recovery to assess rates of relapse and mortality.

ELIGIBILITY:
Inclusion Criteria:

* recovered from moderate acute malnutrition, as defined by mid-upper arm circumference (MUAC) of 11.5-12.4 cm

Exclusion Criteria:

* not permanent resident in vicinity of site
* severe chronic illness
* receiving other supplementary food or participating in other research

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1499 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of children who remain well-nourished (Defined as mid-upper arm circumference (MUAC) > 12.5 cm and without edema) | 12 months
  Defined as mid-upper arm circumference (MUAC) > 12.5 cm and without edema

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Nutrition Project, Blantyre, Malawi

REFERENCES:
- [Derived] Stobaugh HC, Rogers BL, Rosenberg IH, Webb P, Maleta KM, Manary MJ, Trehan I. Children with Poor Linear Growth Are at Risk for Repeated Relapse to Wasting after Recovery from Moderate Acute Malnutrition. J Nutr. 2018 Jun 1;148(6):974-979. doi: 10.1093/jn/nxy033. PMID 29726948
- [Derived] Stobaugh HC, Bollinger LB, Adams SE, Crocker AH, Grise JB, Kennedy JA, Thakwalakwa C, Maleta KM, Dietzen DJ, Manary MJ, Trehan I. Effect of a package of health and nutrition services on sustained recovery in children after moderate acute malnutrition and factors related to sustaining recovery: a cluster-randomized trial. Am J Clin Nutr. 2017 Aug;106(2):657-666. doi: 10.3945/ajcn.116.149799. Epub 2017 Jun 14. PMID 28615258